CLINICAL TRIAL: NCT03957421
Title: Underwater Activity Compared to Land-based Activity for Individuals With Stroke
Brief Title: Aquatic Exercise and Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Methodist University, North Carolina (Other)
Responsible Party: Principal Investigator, Stacia Hall, Assistant Professor of Physical Therapy, Methodist University, North Carolina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5/14/2019 Stroke
Record Dates: First submitted 2019-05-14; First posted 2019-05-21 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Aquatic exercise is more beneficial than land based exercise (Experimental): use of aquatic exercise will be evaluated for individuals with stroke
  Interventions: Other: aquatic exercise, land based exercise

INTERVENTIONS:
Other: aquatic exercise, land based exercise — general warm up and cool down. general exercises and treadmill training at self-selected intensity.

SUMMARY:
To determine the impact of underwater vs. land based exercise and/or gait training on functional mobility for patients with stroke.

DETAILED DESCRIPTION:
Subjects will be recruited via convenience sampling from the Methodist University community and local area. Additionally contacts from medical clinics may be contacted for recruitment of participants. Once individuals have been identified, they will be informed of inclusion and exclusion criteria to be assessed for appropriateness for the project. Informed consent will be provided to participants prior to start.

Inclusion criteria consists of having a stroke and being able to walk 20 meters without a lower extremity orthotic. If participant's have significant fear of water, seizures, incontinence with bowel or bladder, open wounds, infections such as UTI or fever, tracheostomy, nasogastric or gastronomy tube, colostomy, uncontrolled hypertension, skin rash, hard cast due to fracture, isolation precautions, IV or indwelling catheters, uncontrolled agitation, require use of continuous supplemental oxygen, or allergies to chemicals used in a pool, they will not be placed in the underwater groups.

Demographic survey will be provided and filled out prior to the start of data collection.

As physical therapy exercise is within the scope of Physical Therapy Practice and in the state of North Carolina Physical Therapists have direct access to practice without a physician clearance, participants will be assessed using baseline testing (please see below) to ensure medical stability for participation in exercise. Furthermore, participants will be asked if they have been cleared by a physician prior to beginning in exercise (please see consent survey). If individuals evaluated by the supervising physical therapist are deemed to need additional medical clearance from their physician, they will be asked to attain a note from the physician stating they are clear to participate in exercise.

Baseline testing: Participants will complete a basic physical therapy examination consisting of vitals assessment (heart rate, blood pressure, oxygen saturation, rate of perceived exertion and respiratory rate), anthropometric measurements, posture, range of motion, strength testing and use of the following outcome measures to assess self-perception of stroke impact, balance and gait: 4-square step test (FSST), Timed Up and Go (TUG), Dynamic Gait Index (DGI), Romberg, Sharpened Romberg and Single Limb Stance (SLS). Additionally, gait characteristics will be measured using the GAITRite System.

ELIGIBILITY:
Inclusion Criteria:

* Stroke
* Able to walk 20 meters without a lower extremity orthotic.

Exclusion Criteria:

* Significant fear of water
* Seizures
* Incontinence with bowel or bladder
* Open wounds
* Infections such as UTI or fever
* Tracheostomy, nasogastric or gastronomy tube
* Colostomy
* Uncontrolled hypertension
* Skin rash
* Hard cast due to fracture
* Isolation precautions
* IV or indwelling catheters
* Uncontrolled agitation
* Require use of continuous supplemental oxygen
* Allergies to chemicals used in a pool

Max Age: 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2019-01-11 (Actual); Primary Completion 2020-01-11 (Actual); Study Completion 2020-01-11 (Actual)

PRIMARY OUTCOMES:
Dynamic Gait Index | 12 weeks
  8 item gait and balance measure looking at fall risk. participants are scored on a 0-3 scale. 19/24 indicates fall risk.

SECONDARY OUTCOMES:
Romberg | 12 weeks.
  Balance test with standing feet together eyes open and eyes closed for up to 30 seconds on 3 trials
Sharpened Romberg | 12 weeks
  Balance test with standing feet one in front of the other eyes open and eyes closed for up to 30 seconds on 3 trials. repeated with each foot in front
Single limb stance | 12 weeks
  balance test with standing on one leg for up to 30 seconds bilaterally for a total of 3 trails
4-square step test | 12 weeks
  balance test looking at the ability to walk in a square with stepping over obstacles and changing directions. participants are timed for how fast they can place each foot in each square and back for 1 round. greater than 15 seconds indicates fall risk.
Timed Up and Go | 12 weeks.
  Balance test for functional mobility. person starts sitting in a chair, when instructed person stands, walks 10 feet turns around, walks back to the chair and sits down. person is timed for 2 trials. second trial is scored.

CONTACTS AND LOCATIONS:
Locations (1):
- Methodist Universtiy, Fayetteville, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No